CLINICAL TRIAL: NCT02288130
Title: Ulipristal Versus Gonadotropin-releasing Hormone Agonists Prior to Laparoscopic Myomectomy: a Double Blind Randomized Controlled Trial
Brief Title: Ulipristal vs. GnRHa Prior to Laparoscopic Myomectomy
Acronym: MYOMEX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, I. de Milliano, MD, MD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014.421
Record Dates: First submitted 2014-11-06; First posted 2014-11-11 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — Leuprolide; ulipristal; ulipristal acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- GnRHa and placebo tablets (Active Comparator): 11.25 mg Leuproreline injections at the onset of pretreatment with placebo tablets (once daily)
  Interventions: Drug: GnRHa
- Ulipristal (Active Comparator): Three months of Ulipristal 5 mg once daily combined with a single saline injection at the onset of pretreatment (produced as placebo of Leuproreline)
  Interventions: Drug: Ulipristal
- Control (No Intervention): No pre-treatment prior to laparoscopic myomectomy

INTERVENTIONS:
Drug: GnRHa
  Other Names: Lucrin
  Arms: GnRHa and placebo tablets
Drug: Ulipristal
  Other Names: Esmya
  Arms: Ulipristal

SUMMARY:
Rationale: Laparoscopic myomectomy is increasingly performed over laparotomic myomectomy, because of the many benefits for the patient in terms of pain, hospital stay and recovery. In order to increase the success rate of a laparoscopic procedure pre-treatment to decrease the volume might be beneficial. Gonadotropin-releasing hormone agonists (GnRHa) are used for this purpose with good results in terms of volume reduction, but sometimes resulting in loss of distinction of the right surgical planes. Ulipristal is a new pre-operative treatment option for symptomatic fibroids, which has demonstrated good results in terms of volume reduction. The effect on cleavage planes is unknown. This study is performed to evaluate if Ulipristal is as effective as GnRHa in terms of surgical outcome.

Objective: to investigate if Ulipristal is non-inferior to GnRH in terms of intra-operative blood-loss (primary outcome), surgical time, surgical ease, complications, quality of life and costs.

Study design: Double blind randomized controlled multi-center trial. Study population: Premenopausal women in whom a maximum of 2 symptomatic intramural fibroids between 5 and 12 cm in diameter will be removed. Fibroid types 3, 4, 5, 6 and 2-5 will be included.

Intervention: Three months of Ulipristal 5 mg once daily combined with a single saline injection at the onset of pretreatment (produced as placebo of Leuproreline) or (comparison) 11.25 mg Leuproreline injections at the onset of pretreatment with placebo tablets (once daily) .

Methods: Within 1 month after pre-treatment patients will undergo a laparoscopic myomectomy by experienced surgeons. Operative characteristics will be recorded prospectively. Follow up will be 6 months after surgery mainly for quality of life assessment. A cost utility analysis will be conducted alongside the trial.

Main study parameters/endpoints: Ulipristal is non-inferior to GnRHa in terms of blood loss during surgery when the average difference between the two groups is below 150 ml (standard deviation 250 ml).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Both Ulipristal and GnRHa have been registered for this indication. Safety has been tested and no specific risks apply.

ELIGIBILITY:
Inclusion Criteria:

Women visiting the gynecological outpatient department with symptomatic fibroids will be screened for eligibility. In order to be eligible to participate in this trial, a subject must meet all of the following criteria:

* provide written consent prior to any study related procedures
* pre-menopausal
* a planned resection of a maximum of 2 FIGO (PALM-COEIN classification) type 3, 4, 5, 6 or 2-5 fibroids of >5 cm
* the(se) fibroid(s) should be between 5 and 12 cm (maximum diameter)
* other fibroids should be small (<2 cm), not clinically relevant, or not resectable (e.g. difficult position), or type 7 (any size)
* eligible for laparoscopic myomectomy

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this trial:

* Current pregnancy
* (suspicion of) malignancy
* any type 0-2 fibroids smaller than 5 cm
* more than 2 type 3-6 fibroids > 5 cm that need to be removed (except type 7 fibroids of any size)
* use of any hormonal agents and not willing to discontinue their use
* use of anticoagulants
* coagulopathy
* Use of NSAIDs impacting bleeding before surgery
* Contraindication to laparoscopy procedure or causes of complications (multiple laparotomies, frozen pelvis, severe endometriosis)
* allergy to leuprolide acetate/comparable nonapeptides or Ulipristal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-07 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Blood loss during surgery | Reported directly after surgery
  Ulipristal is non-inferior to GnRHa in terms of blood loss during surgery when the average difference between the two groups is below 150 ml (standard deviation 250 ml)

CONTACTS AND LOCATIONS:
Overall Officials: Wouter Hehenkamp, PhD, Study Chair — Amsterdam UMC, location VUmc
Locations (9):
- Netherlands (9):
  - Flevoziekenhuis, Almere Stad
  - Onze Lieve Vrouwen Gasthuis, Amsterdam
  - Sint Lucas Andreas Ziekenhuis, Amsterdam
  - VU medical center, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - Spaarne Gasthuis, Haarlem
  - Radboud University Medical Center, Nijmegen
  - Maasstad ziekenhuis, Rotterdam
  - Maxima Medisch Centrum, Veldhoven